CLINICAL TRIAL: NCT04839458
Title: Investigation of the Effect of Scan Delay on the Measurement of Dental Prescale II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 202102052RINA
Record Dates: First submitted 2021-04-05; First posted 2021-04-09 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2022-06

CONDITIONS: Bite Force; Scan Delay
Keywords: Dental Prescale II,Scan Delay

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dental Prescale II used (Experimental)
  Interventions: Device: Dental Prescale II

INTERVENTIONS:
Device: Dental Prescale II — The participant will bite Dental Prescale II for about 3 seconds, using a force for " chewing beef ". And the Dental Prescale II will be taken out from the mouth. Then the trial is end.

SUMMARY:
Dental Prescale II (GC Corp., Tokyo) is a pressure sensitive sheet for occlusal force measurement. According to the instruction, the patient need to bite the sheet for about 3 seconds and then the sheet will be scanned. But the delay response of coloring agent will influence the data collected and was noticed in vitro. To have a standard procedure, we need to know the time for scanning. This study will scan the sheet up to 2 hours and try to find the relation between the time the sheet scanned and the data collected.

ELIGIBILITY:
1. Inclusive criteria:

   * full dentition except third molar
   * healthy periodontal condition
   * can sign consent
2. Exclusive criteria:

   * history of temporomandibular disorders

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
The relation between occlusal force and scanning time | immediately after the intervention
  After Dental Prescale II is used and cleaned, the first time of scanning will be defined as 0 min. The pressure sensitive sheet will be scanned every minute during 0~15 minutes, and at 30, 60, 90 and 120 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: TongMei Wang Wang, PHD, Principal Investigator — School of Dentistry, National Taiwan University College of Medicine.
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng District, Taiwan